CLINICAL TRIAL: NCT05747820
Title: Observational Study for Multiparametric Assessment of Cardiac Congestion in Outpatient Worsening Heart Failure (EVOLUTION)
Brief Title: Multiparametric Assessment of Cardiac Congestion in Outpatient Worsening Heart Failure
Acronym: EVOLUTION
Status: Completed | Type: Observational
Sponsor: Corteria Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CHF202102
Record Dates: First submitted 2023-02-08; First posted 2023-02-28 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Heart Decompensation
Keywords: Worsening Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (plasma) and urine samples for central laboratory assessment will be taken at Visits 1, and Visit 5. Sample aliquots will be stored frozen locally until shipped for longer-term storage and analysis. Unused samples will be discarded within 7 years after the study's completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — This is an observational study designed to assess the evolution of multiple markers of congestion over 4 weeks after a WHF event treated in an outpatient unit

SUMMARY:
This observational study is conducted to assess the evolution of multiple markers of congestion over 4 weeks after a worsening heart failure (WHF) event treated in an outpatient unit

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, observational study designed to assess the evolution of multiple markers (physical, echocardiographic, and biomarkers) of congestion in 40 patients with chronic heart failure (CHF) treated over 4 weeks with 40 to 120 mg daily oral furosemide after an event of WHF treated in an outpatient unit. Patients at selected centers may participate in a telemetry ancillary study, in which real-time, continuous, non-invasive measurements of physiologic parameters of heart failure will be obtained through use of a wearable medical telemetry device.

Approximately 40 patients with CHF with reduced or mildly reduced left ventricular ejection fraction (EF < 50%) who had an admission for WHF in the preceding 1-12 months and who develop symptoms of WHF over the week before presentation to an outpatient clinic will be enrolled. Patients will attend five outpatient visits over the course of 4 weeks.

At each visit, the patient's vital signs will be measured, clinical assessments (NYHA class, jugular vein distension, peripheral edema score, pulmonary rales) will be performed, and blood samples for central assays will be obtained. Detailed echocardiographic examination will be performed prior to enrolment in the first visit and at Visit 5.

Biomarkers related to cardiac and renal function will be measured in blood and urine samples at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 and < 80 years of age.
2. Previous documented hospital admission for HF between 12 months and 1 month prior to Screening.
3. Ambulatory patients with a diagnosis of stable NYHA class II - III HF with left ventricular ejection fraction <50%, who experience a worsening of heart failure (WHF), with worsening signs and/or symptoms of heart failure requiring institution or up titration of loop diuretic therapy, in the week preceding their visit to the outpatient HF clinic and with at the time of Screening:

   1. Dyspnea and at least one symptom of congestion (rales, orthopnea, peripheral oedema)
   2. Imaging confirmation of congestion as defined by either pulmonary congestion on chest X-ray or at least 2 B-lines by lung ultrasound.
4. Stable oral doses of ACEi, ARB or ARNi, beta-blocker, mineralocorticoid antagonist (MRA), and SGLT2i for > 1 month prior to screening.
5. An increase in the prescribed oral loop diuretic dose up to 120 mg daily furosemide or equivalent*for the treatment of the WHF event.
6. Biomarker profile suggestive of significant HF inclusive of NT-proBNP ≥1500 pg/ml, and elevated TnT from 15 ng/L (0.015 mcg/L) to 150 ng/L (0.15 mcg/L) or equivalent TnI using ultrasensitive assay.
7. Mild to moderate renal impairment (eGFR by the simplified MDRD formula of >30 and <60 ml/min/1.73 m2).
8. Written informed consent to participate in the study.
9. Ability to comply with all study requirements, without major morbidities compromising the patient's ability to participate and understand the study for 90 days.

Exclusion Criteria:

1. Significant pulmonary disease contributing substantially to the patients' dyspnea such as FEV1< 1 liter or need for chronic steroid therapy.
2. Myocardial infarction, unstable angina, ICD or CRT implantation, or cardiac surgery, including percutaneous transluminal coronary intervention, within past 3 months.
3. History of heart transplant or on a transplant list or using or planned to be implanted with a ventricular assist device.
4. Significant uncontrolled arrythmia such as atrial fibrillation with a persistent heart rate > 120 beast/minute, any bradyarrhythmia with a persistent heart rate < 50 beats/min, sustained supraventricular tachycardia, any evidence of tri-fascicular block by ECG.
5. Sustained ventricular arrhythmia with syncopal episodes within past 3 months that is untreated.
6. Presence of any hemodynamically moderate or severe valvular stenosis or regurgitation, except for moderate mitral or tricuspid regurgitation secondary to left ventricular dilatation. Presence of hemodynamically significant obstructive lesions of left ventricular outflow tract.
7. Stroke or TIA within the past 3 months.
8. Primary or alcoholic liver disease considered to be life threatening.
9. Any episode of symptomatic hypotension within 3 months prior to screening.
10. Coagulation or bleeding disorder.
11. Systolic blood pressure < 100 mmHg or >180 mmHg.
12. Serum sodium > 146 mEq/L (146 mmol/L) or <135 mEq/L
13. Serum potassium > 5.2 mEq/L (5.2 mmol/L) or < 3.5 mEq/L (3.5 mmol/ L).
14. Ultrafiltration or dialysis within 3 months prior to Screening.
15. Hypersensitivity to furosemide.
16. History or presence of any other diseases (i.e. including malignancies) with a life expectancy of < 3 months.
17. Participation in any CHF trial or any investigational drug or device study within the 30 days prior to Screening.
18. History of noncompliance to medical regimens and patients who are considered potentially unreliable.
19. Pregnant or nursing (lactating) women.
20. Active infection based on abnormal temperature and/or elevated WBC count.
21. Any evidence of COVID -19 infection
22. Hemoglobin <8 g/L or receipt of blood transfusion within 3 months prior to Screening.
23. Contraindication to the use of the wrist-worn telemetry device: skin problem or wound in the wrist area, inclusive of tattoos.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 40 adult male and female patients with a diagnosis of HFrEF (EF<40%) and HFmrEF (EF >40 < 50%) who had a hospital admission for HF within 1 to12 months prior to screening and developed worsening symptoms of HF during the week prior to presentation to an outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Change in E/e' ratio | Screening (Visit 1) and week 4 (beginning of Visit 5).
  Change in E/e' ratio, measured on echocardiography
Changes in Left Ventricular End-Diastolic Diameter (LVEDD) | From screening to 4 weeks
  Changes in LVEDD measured on echocardiography from screening to Week 4
Changes in Left Ventricular End-Systolic Diameter (LVESD) | From screening to 4 weeks
  Changes in LVESD measured on echocardiography from screening to Week 4
Changes in Left Ventricular End-Diastolic Volume (LVEDV) | From screening to 4 weeks
  Changes in LVEDV measured on echocardiography from screening to Week 4
Changes in Left Ventricular End-Systolic Volume (LVESV) | From screening to 4 weeks
  Changes in LVESV measured on echocardiography from screening to Week 4
Changes in Left Ventricular Ejection Fraction (LVEF) | From screening to 4 weeks
  Changes in LVEF measured on echocardiography from screening to Week 4
Changes in mitral E-velocity | From screening to 4 weeks
  Changes in mitral E-velocity measured on echocardiography from screening to Week 4
Changes in mitral A-velocity | From screening to 4 weeks
  Changes in mitral A-velocity measured on echocardiography from screening to Week 4
Changes in E' velocity | From screening to 4 weeks
  Changes in E' velocity measured on echocardiography from screening to Week 4
Changes in Right Ventricular Systolic Pressure (RVSP) | From screening to 4 weeks
  Changes in RVSP measured on echocardiography from screening to Week 4
Changes in Tricuspid Annular Pulmonary Systolic Excursion (TAPSE) | From screening to 4 weeks
  Changes in TAPSE measured on echocardiography from screening to Week 4
Changes in S' velocity | From screening to 4 weeks
  Changes in S' velocity measured on echocardiography from screening to Week 4
Changes in Inferior Vena Cava (IVC) diameter | From screening to 4 weeks
  Changes in IVC (minimum and maximum) measured on echocardiography from screening to Week 4
Changes in Left Atrium (LA) surface | From screening to 4 weeks
  Changes in LA surface measured on echocardiography from screening to Week 4
Changes in Right Atrium (RA) surface | From screening to 4 weeks
  Changes in RA surface measured on echocardiography from screening to Week 4
Changes in patient-reported dyspnea | From screening to 4 weeks
  Weekly changes in patient-reported dyspnea
Changes in clinically-assessed jugular venous pulse | From screening to 4 weeks
  Weekly changes in clinically-assessed jugular venous pulse
Changes in clinically-assessed peripheral edema | From screening to 4 weeks
  Weekly changes in peripheral edema
Changes in estimated Glomerular Filtration Rate (eGFR) | From screening to 4 weeks
  Changes in eGFR between screening, Week 2 and Week 4 visit.
Changes in serum creatinine | From screening to 4 weeks
  Changes in serum creatinine between screening, Week 2 and Week 4 visit.
Changes in NT-proBNP | From screening to 4 weeks
  Changes in NTproBNP between screening, Week 2 and Week 4 visit.
Changes in high sensitivity Troponin T (HsTnT) | From screening to 4 weeks
  Changes in HsTnT between screening, Week 2 and Week 4 visit.
Changes in Kansas City Cardiomyopathy Questionnaire (KCCQ)-12 | From screening to 4 weeks
  Changes in KCCQ-12 inclusive of total symptoms score and sub scores from screening to Week 4
Weekly changes in telemetered parameters in patients wearing the wrist-worn device (Philips Health Band) | From screening to 4 weeks
  Weekly changes in activity in those patients wearing the wrist-worn device (Philips Health Band)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, MD, Principal Investigator — Hôpitaux Universitaires Saint-Louis-Lariboisière, University Paris Diderot, Inserm 942
Locations (4):
- Armenia (2):
  - Institute of Cardiology Levon Hovhannisyan, Yerevan
  - Erebuni Medical Center, Yerevan
- Bosnia and Herzegovina (2):
  - Health Institution Medico Laser, Cardiology ward, Banja Luka
  - Universty Clinical Hospital Mostar, Clinic for Internal diseases with dyalisis center, Clinical ward for cardiology, Mostar

IPD SHARING:
Plan to Share IPD: No